CLINICAL TRIAL: NCT02610153
Title: A Prospective Observational Study Assessing the Management of Anticoagulation With Vitamin K Antagonists in Patients With Nonvalvular Atrial Fibrillation Treated in Cardiology Practices
Brief Title: Subtherapeutic INR Levels in Patients With AVK: Incidence, Associated Factors, Prognosis and Control Strategies
Acronym: SULTAN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17943
Record Dates: First submitted 2015-10-20; First posted 2015-11-20 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — acarboxyprothrombin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Adult patients, diagnosed with no-valvular atrial fibrillation and who have recently initiated or are going to initiate VKA treatment, that attend the Cardiology Units
  Interventions: Drug: Vitamin K Antagonist

INTERVENTIONS:
Drug: Vitamin K Antagonist — The vitamin K antagonists exert their anticoagulant effect through inhibition of the enzyme complex of vitamin K epoxide reductase subunit 1 with subsequent reduction of the gamma-carboxylation of certain glutamic acid molecules endpoints located on factors coagulation II (prothrombin), VII, IX and X and protein C or its cofactor protein S. This gamma-carboxylation has a significant bearing on the interaction of coagulation factors referenced with calcium ions. Without this reaction, blood clotting cannot be initiated. The dose must be adjusted to each patient at baseline and after regular basis, since the sensitivity to anticoagulants varies between individuals and can also vary throughout the treatment. For this, the Prothrombin Time (PT) is used and standardized ratio called International Normalised Ratio (INR).

SUMMARY:
This prospective observational study is to assess the predictive factors of poor control of international normalized ratio (INR) to determine the treatment strategies received by patients with a poor control of INR in real-life clinical practice and to explore the effectiveness and safety of these strategies in patients with non-valvular atrial fibrillation who start vitamin K antagonist (VKA) treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Patients with a diagnosis of nonvalvular atrial fibrillation according to the criteria of the Spanish Agency of Medicines and Medical Devices (AEMPS) (2013) who are treated in cardiology practices.
* Patients about to start treatment with a vitamin K antagonist or who are in the first two months of treatment.
* Patients for whom access to at least 80% of INR tests performed during treatment with vitamin K antagonists is expected to be available.
* Patients with the mental and physical capacity to complete the study questionnaires and give their informed consent to participate in the study.

Exclusion Criteria:

* Patients with mitral stenosis or another significant valve disease for which specific treatment is scheduled or has already been performed (prosthesis or valvuloplasty).
* Patients hospitalised at the time of inclusion in the study.
* Patients with a life expectancy of less than 13 months.
* Patients who are participating in a clinical trial.
* Patients receiving double antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-valvular atrial fibrillation who are going to start vitamine K antagonist treatment or have started over the previous two months and that attend the Cardiology Units at Spanish hospitals (as outpatients).
Sampling Method: Non-Probability Sample
Enrollment: 1013 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
International Normalized Ratio (INR) Time in Therapeutic Range (TTR) | Up to 24 months
  Percentage of time within an INR range of 2-3 estimated using the Rosendaal method

SECONDARY OUTCOMES:
Baseline thromboembolic risk based on the CHADS2 scale | Baseline
  CHADS2: Cardiac failure, Hypertension, Age, Diabetes, Stroke
Baseline thromboembolic risk based on the CHA2DS2-VASc scale | Baseline
  CHA2DS2-VASc:Cardiac failure, Hypertension, Age ≥75, Diabetes, Stroke -Vascular disease, Age and sex category
Baseline haemorrhagic risk based on the HAS-BLED scale | Baseline
  HAS-BLED: Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or predisposition, Labile INR, Elderly , Drugs/alcohol
Changes in INR time in therapeutic range | Up to 24 months
  INR time in therapeutic range: percentage of time within an INR range of 2-3 estimated using the Rosendaal method
Patient preferences with regard to anticoagulant treatment based on patients' questionnaires | Up to 12 months
Satisfaction with the anticoagulant treatment based on the Anti-Clot Treatment Scale (ACTS) | Up to 12 months
Adherence to the anticoagulant treatment: Morisky-Green test | Up to 12 months
Number and type of visits by patients to health professionals related to their anticoagulant treatment | Up to 12 months
Number of patients using anticoagulant treatment strategies | Up to 24 months
  Strategies: patients continuing vitamin K antagonists, patients with changes/adjustments to the dose of vitamin K antagonists and patients whose treatment is changed to direct action oral anticoagulants
Number of patients treated according to clinical practice guidelines based on the Spanish Agency of Medicines and Medical Devices (AEMPS) therapeutic positioning report | Up to 24 months
Number of thromboembolic events in patients with inadequate anticoagulation management | Up to 24 months
Number of haemorrhagic events in patients with inadequate anticoagulation management | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Spain